CLINICAL TRIAL: NCT06180928
Title: Short Term Outcome of Metabolic Associated Fatty Liver Disease (MAFLD) in Patients Undergoing Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Essam Mohie Atef Sayed, priniciple investigator, Assiut University
Other Study IDs: MAFLD and bariatric surgery
Record Dates: First submitted 2023-12-03; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Metabolic Associated Fatty Liver Disease; Bariatric Surgery Candidate
Keywords: MAFLD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity has become one of the most critical public health problems in economically developed and developing countries in the world.

Bariatric surgery is an option for obese individuals who fail to achieve suitable weight loss with lifestyle changes and pharmacological methods. Bariatric surgery can help obese individuals achieve recommended weight reduction and thus improve the course of MAFLD. The additional benefits of bariatric surgery include resolution or amelioration of hypertension, hyperlipidemia and type 2 diabetes and reduction of cardiovascular risk and mortality .

The relation between rate of weight loss after bariatric surgeries and the course of the MAFLD not well studied befor ,So we are aiming to assess the outcome of MAFLD ,TSH in patients undergoing Barietric surgeries and if there is significant correlation of steatosis and rate of weight loss among those patients.

DETAILED DESCRIPTION:
Obesity has become one of the most critical public health problems in economically developed and developing countries in the world. It causes metabolic disorders that increase the risk of mortality and morbidity in adulthood. Furthermore, obesity contributes significantly to the pathogenesis of diabetes mellitus, cardiovascular disease, hyperlipidemia, obstructive sleep apnea, and hypertension pathogenesis.

Non-alcoholic fatty liver disease (NAFLD) is defined by macrovesicular steatosis in 5% hepatocytes, in the absence of a secondary cause such as alcohol or drugs. It includes a spectrum of diseases from non-alcoholic fatty liver (NAFL) through to non-alcoholic steatohepatitis (NASH), fibrosis and cirrhosis. The worldwide prevalence of NAFLD is about 25%, ranging from 13% in Africa to 23% in Europe and 32% in the Middle East. Non-alcoholic fatty liver disease (NAFLD) is a recognized complication of obesity.

Recently, it has been proposed to change the name of non-alcoholic fatty liver disease (NAFLD) to Metabolic Associated Fatty Liver Disease (MAFLD) to better reflect the pathophysiology of the disease. MAFLD may better reflect the pathophysiology of this disorder and provides a broad definition for this heterogeneous disorder. The criteria are based on the evidence of hepatic steatosis, plus any of the following three conditions: overweight/ obesity, presence of type 2 diabetes mellitus (T2DM), or evidence of metabolic dysregulation.

Obesity is associated with high TSH levels. Clinical studies have shown a positive correlation between obesity and plasma TSH levels. Furthermore, weight loss in these patients is associated with changes in serum TSH and thyroid hormone levels.

Bariatric surgery is an option for obese individuals who fail to achieve suitable weight loss with lifestyle changes and pharmacological methods. Bariatric surgery can help obese individuals achieve recommended weight reduction and thus improve the course of MAFLD. The additional benefits of bariatric surgery include resolution or amelioration of hypertension, hyperlipidemia and type 2 diabetes and reduction of cardiovascular risk and mortality .

Also The decrease in adipose tissue after bariatric surgery causes changes in plasma fT3, fT4, and TSH levels. obese patients had a decreased thyroid hormone gene expression (especially TSH receptor) in subcutaneous and visceral adipose tissue.

The relation between rate of weight loss after bariatric surgeries and the course of the MAFLD not well studied befor ,So we are aiming to assess the outcome of MAFLD ,TSH in egyption patients undergoing Barietric surgeries and if there is significant correlation of steatosis and rate of weight loss among those patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years old and diagnosed with metabolic associated fatty liver disease and planning to undergo bariatric surgery

Exclusion Criteria:

1. Age below 18 years old.
2. Patients have history of HBV...HCV
3. patients with autoimmune hepatitis
4. Alcoholic patients
5. Drug induced hepatitis
6. Willson Diseaese
7. Haemochromatosis Diseaese

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients more than 18 years old and diagnosed with metabolic associated fatty liver disease and planning to undergo bariatric surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of bariatric surgery in the course of hepatic steatosis among MAFLD patients. | baseline
  fiboscan as A CAP score that falls anywhere between 238 to 260 dB/m represents 11-33% fatty change in the liver. A CAP score that falls anywhere between 260 to 290 dB/m represents 34-66% fatty change in the liver. A CAP score that is 290 dB/m or higher represents over 67% fatty change in the liver
studying effect of weight reduction at the level of TSH | baseline
  Measure the level TSH (mIU/L) in patienta befor and after bariatric surgery incorrolation on weight loss (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Zeinelabdeen Ahmed Sayed, Professor, Study Chair — Assiut University; Ghada AbdelRahman, professor, Study Director — Assiut University; bahaa osman, lecturer, Study Director — Assiut University

REFERENCES:
- [Result] Lin X, Li H. Obesity: Epidemiology, Pathophysiology, and Therapeutics. Front Endocrinol (Lausanne). 2021 Sep 6;12:706978. doi: 10.3389/fendo.2021.706978. eCollection 2021. PMID 34552557
- [Result] Le MH, Yeo YH, Zou B, Barnet S, Henry L, Cheung R, Nguyen MH. Forecasted 2040 global prevalence of nonalcoholic fatty liver disease using hierarchical bayesian approach. Clin Mol Hepatol. 2022 Oct;28(4):841-850. doi: 10.3350/cmh.2022.0239. Epub 2022 Sep 19. PMID 36117442
- [Result] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314
- [Result] Kamal MEEM, Aisha HAA, Fahmy MH, Abosayed AK. The Impact of Laparoscopic Sleeve Gastrectomy on Thyroid Functions in Egyptian Patients with Obesity. J Gastrointest Surg. 2023 Jul;27(7):1345-1352. doi: 10.1007/s11605-023-05662-4. Epub 2023 Apr 5. PMID 37020159
- [Result] Diemieszczyk I, Wozniewska P, Golaszewski P, Drygalski K, Nadolny K, Ladny JR, Razak Hady H. Does weight loss after laparoscopic sleeve gastrectomy contribute to reduction in blood pressure? Pol Arch Intern Med. 2021 Aug 30;131(7-8):693-700. doi: 10.20452/pamw.16023. Epub 2021 Jun 2. PMID 34075736
- [Result] Nannipieri M, Cecchetti F, Anselmino M, Mancini E, Marchetti G, Bonotti A, Baldi S, Solito B, Giannetti M, Pinchera A, Santini F, Ferrannini E. Pattern of expression of adiponectin receptors in human liver and its relation to nonalcoholic steatohepatitis. Obes Surg. 2009 Apr;19(4):467-74. doi: 10.1007/s11695-008-9701-x. Epub 2008 Oct 16. PMID 18923878
- [Result] Lassailly G, Caiazzo R, Buob D, Pigeyre M, Verkindt H, Labreuche J, Raverdy V, Leteurtre E, Dharancy S, Louvet A, Romon M, Duhamel A, Pattou F, Mathurin P. Bariatric Surgery Reduces Features of Nonalcoholic Steatohepatitis in Morbidly Obese Patients. Gastroenterology. 2015 Aug;149(2):379-88; quiz e15-6. doi: 10.1053/j.gastro.2015.04.014. Epub 2015 Apr 25. PMID 25917783
- [Result] Pasquali R, Casanueva F, Haluzik M, van Hulsteijn L, Ledoux S, Monteiro MP, Salvador J, Santini F, Toplak H, Dekkers OM. European Society of Endocrinology Clinical Practice Guideline: Endocrine work-up in obesity. Eur J Endocrinol. 2020 Jan;182(1):G1-G32. doi: 10.1530/EJE-19-0893. PMID 31855556